CLINICAL TRIAL: NCT04955548
Title: A Clinical Translational Study on Repairing Articular Cartilage Injury With Autologous Adipose Gel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2020311
Record Dates: First submitted 2021-06-25; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Articular Cartilage Defects

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arthroscopic microfracture with autologous adipose gel (Experimental): The experimental group will be treated with arthroscopic microfracture with autologous adipose gel.
  Interventions: Procedure: arthroscopic micro-fracture with autologous adipose gel
- arthroscopic microfracture (Active Comparator): The control group will be treated with arthroscopic microfracture.
  Interventions: Procedure: arthroscopic micro-fracture

INTERVENTIONS:
Procedure: arthroscopic micro-fracture with autologous adipose gel — Fully cut the adipose tissue taken out under the arthroscopy, transfer the cut adipose tissue to a syringe connected with a double pass, push back and forth through the syringe to physically emulsify the adipose, and centrifuge to obtain the autologous adipose gel, and inject it into the lesion
  Arms: arthroscopic microfracture with autologous adipose gel
Procedure: arthroscopic micro-fracture — Surgeons routinely perform international standard micro-fracture surgery to repair cartilage damage
  Arms: arthroscopic microfracture

SUMMARY:
66 articular cartilage injury diseases patients were divided into two groups as 1:1. The test group will be treated with arthroscopic micro-fracture with autologous adipose gel, and the control group will be treated with arthroscopic micro-fracture. Postoperative MRI evaluation, Lysholm score, IKDC score, Tegner score, and VAS score will be used as the treatment validity evaluation index, at the same time testing blood routine, blood biochemistry, urine routine, CRP, electrocardiogram and other laboratory tests and recording the occurrence of adverse events.

DETAILED DESCRIPTION:
In this study, 66 patients who were clinically diagnosed as articular cartilage injury diseases were divided into test group and control group according to the ratio of 1:1. The test group will be treated with arthroscopic micro-fracture with autologous adipose gel, and the control group will be treated with arthroscopic micro-fracture. Postoperative MRI evaluation, Lysholm score, IKDC score, Tegner score, and VAS score will be used as the treatment validity evaluation index, at the same time testing blood routine, blood biochemistry, urine routine, CRP, electrocardiogram and other laboratory tests and recording the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old and ≤50 years old, male or female patients
2. Patients with knee articular cartilage defect area ≥2cm2 and ≤8cm2, who can undergo microfracture surgery, no surgical contraindications
3. Patients voluntarily participate in clinical trials, sign an informed consent form, and be able to cooperate with clinical follow-up

Exclusion Criteria:

1. Participants in clinical trials of other drugs or medical devices in the past 6 months
2. Unable to accept autologous fat glue due to religion, ethnicity, etc.
3. Injury area <2 cm2 or >8cm2 or lack of normal cartilage tissue surrounding the injury
4. Those with compound multiple ligament injuries
5. Those with systemic immune diseases or systemic or local infections
6. Those with joint fibrosis, joint ankylosis, and obvious limitation of movement
7. People with moderate to severe osteoarthritis
8. Those who have contraindications to MRI examination
9. Patients with hemophilia
10. People whose general condition cannot tolerate surgery
11. Women who are pregnant or planning to become pregnant and women who are breastfeeding
12. Mental abnormalities and no behavioral autonomy
13. Other circumstances in which the doctor judges that he cannot participate in the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessing a change of MRI Evaluation of Articular Cartilage Injury after Repair | Knee MRI examinations were performed on patients baseline, 5 days, 90 days, 180 days, and 365 days after operation.
  Assessing a change of postoperative MRI evaluation with autologous fat glue combined with micro-fracture treatment or micro-fracture treatment articular cartilage injury

SECONDARY OUTCOMES:
Lysholm score | Lysholm score was tested for the two groups of patients' baseline, 5 days, 90 days, 180 days, and 365 days after operation.
  Assessing a change of Lysholm score between two groups of patients
IKDC score | IKDC score was tested for the two groups of patients' baseline, 5 days, 90 days, 180 days, and 365 days after operation.
  Assessing a change of IKDC score between two groups of patients
Tegner score | Tegner score was tested for the two groups of patients' baseline, 5 days, 90 days, 180 days, and 365 days after operation.
  Assessing a change of Tegner score between two groups of patients
VAS score | VAS score was tested for the two groups of patients' baseline, 5 days, 90 days, 180 days, and 365 days after operation.
  Assessing a change of VAS score between two groups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Yingfang Ao, Prof., Principal Investigator — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing Key Laboratory of Sports Injuries， Beijing, China, Beijing, Beijing Municipality, China